CLINICAL TRIAL: NCT01541969
Title: Systematic Evaluation of the Acoustic CR ® Neuromodulation Treatment for Tinnitus
Brief Title: Evaluation of the CR Neuromodulation Treatment for Tinnitus
Acronym: RESET2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: University of Nottingham (Other); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11IH006
Record Dates: First submitted 2012-02-24; First posted 2012-03-01 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2015-05

CONDITIONS: Tinnitus
Keywords: Ear; Hearing
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CR Neuromodulation (Experimental): Adaptive NeuroModulation (ANM) T30 CR® Neurostimulator device. Participants receive the intervention according to the manufacturer/funder training given to the study team.
  Interventions: Device: CR Neuromodulation
- Tinnitus masking (Active Comparator): Participants will receive the same Adaptive NeuroModulation (ANM) T30 CR® Neurostimulator device, but it will NOT be programmed according to the therapeutic algorithm (0-12 weeks).
  Interventions: Device: Tinnitus masking

INTERVENTIONS:
Device: CR Neuromodulation — Ear level device which delivers patterned sound stimulation.
  The experimental arm will use the device fitted according to audiologist training given by the manufacturer/funder. An individually specified sound stimulation algorithm is hypothesised to interrupt tinnitus generating activity in the brain. For the first 12 weeks participants will be asked to wear the device every day for 6 hours, and in blocks of time not less than 1 hour. After 12 weeks participants will be unblinded and continue with the same experimental intervention. In weeks 13-36 participants will be asked to wear the device every day for 4 hours, in continuous blocks of at least 1 hour.
  Other Names: Acoustic Coordinated Reset Neuromodualtion
  Arms: CR Neuromodulation
Device: Tinnitus masking — The active comparator uses the same ear level device and also delivers patterned sound but the stimulus will be determined according to an algorithm predicted not to break up tinnitus generating activity in the brain. It may have a masking effect. For the first 12 weeks participants will be asked to wear the device every day for 6 hours, and in blocks of time not less than 1 hour. After 12 weeks, the participants will be unblinded and the device algorithm will be reprogrammed in the same way as the experimental intervention. In weeks 13-24 participants will be asked to wear the device for 6 hours per day, in continuous blocks of at least 1 hour. In weeks 25-36 they will be asked to continue using the device every day for 4 hours, in continuous blocks of at least 1 hour.
  Other Names: Tinnitus masking only (by CR Neuromodulation device)
  Arms: Tinnitus masking

SUMMARY:
The purpose of this study is to determine whether a new device delivering a sound-based intervention (termed acoustic coordinated reset neuromodulation) has significant clinical benefit for people with intrusive tinnitus. It is hypothesised that the particular pattern of sound stimulation delivered by the device acts to break up patterns of synchronous nerve firing in the brain that may be responsible for the sensation of tinnitus. We will also measure brain activity in a subset of participants to determine if the intervention results in changes in brainwave activity.

DETAILED DESCRIPTION:
Tinnitus affects a large number of people in the UK population but is a poorly understood disorder with no form of treatment that benefits everyone. One theory about tinnitus is that it is caused by altered patterns of synchronous nerve firing in the brains hearing centres. It is believed that conditions such as hearing loss lead to changes in how areas of the brain responsible for hearing are 'wired up' causing large areas of the brain to fire at the same time; this is believed to be a mechanism responsible for the sensation of tinnitus. Research suggests that this type of synchronous activity may be interrupted by presenting very specific sequences of sounds to the ears over several months. If sound stimulation can be used to break up patterns of synchronous activity in the hearing brain, then it is argued that it should also be effective in treating tinnitus. The German company ANM have patented a very specific algorithm of sound simulation that is delivered via headphones from a pocket-sized device. This treatment is currently being marketed by the private healthcare sector in Germany and very recently in the UK. The purpose of this study is to independently test the effects of this new therapy on tinnitus severity and related brain activity. We will gather information using questionnaires and listening tests, and make recording of electrical brain activity using electroencephalography (EEG).

ELIGIBILITY:
Inclusion Criteria:

* Pure tone average <60 dB HL in the ear where tinnitus is perceived
* Must be able to hear all stimulation tones presented by the device
* Chronic subjective tinnitus for more than 3 months
* Dominant tinnitus frequency measured between 0.2 and 10 kHz
* At least mild tinnitus score on the Tinnitus Handicap Inventory
* Willing to wear the device for 4-6 hours daily during the trial
* Sufficient command of English language to read, understand and complete the questionnaires
* Able and willing to give informed consent

Exclusion Criteria:

* Objective tinnitus, Meniere's disease, craniomandibular induced Tinnitus
* Pulsatile tinnitus
* Intermittent tinnitus
* Severe anxiety
* Severe depression
* Catastrophic tinnitus
* Hearing-aids wearers for less than 9 months
* Hearing-aid wearers with audiological adjustments within last 3 months
* Absolute thresholds > 70 dB on individual frequencies up to 8 kHz (unable to sufficiently hear the stimulus)
* Taking part in another trial during the last 30 days before study start
* The individually tailored training stimulus is uncomfortable or not acceptable to the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Hall, PhD, Study Director — NIHR Nottingham Hearing Biomedical Research Unit, Unviersity of Nottingham; Derek J Hoare, PhD, Principal Investigator — NIHR Nottingham Hearing Biomedical Research Unit, University of Nottingham; David McAlpine, PhD, Principal Investigator — University College London, Ear Institute
Locations (2):
- United Kingdom (2):
  - University College London Ear Institute, London
  - NIHR Nottingham Hearing Biomedical Research Unit, University of Nottingham, Nottingham

REFERENCES:
- [Background] Hoare DJ, Edmondson-Jones M, Gander PE, Hall DA. Agreement and reliability of tinnitus loudness matching and pitch likeness rating. PLoS One. 2014 Dec 5;9(12):e114553. doi: 10.1371/journal.pone.0114553. eCollection 2014. PMID 25478690
- [Background] Hoare DJ, Pierzycki RH, Thomas H, McAlpine D, Hall DA. Evaluation of the acoustic coordinated reset (CR(R)) neuromodulation therapy for tinnitus: study protocol for a double-blind randomized placebo-controlled trial. Trials. 2013 Jul 10;14:207. doi: 10.1186/1745-6215-14-207. PMID 23842505
- [Background] Fackrell K, Hall DA, Barry JG, Hoare DJ. Psychometric properties of the Tinnitus Functional Index (TFI): Assessment in a UK research volunteer population. Hear Res. 2016 May;335:220-235. doi: 10.1016/j.heares.2015.09.009. Epub 2015 Sep 28. PMID 26415998
- [Background] Pierzycki RH, McNamara AJ, Hoare DJ, Hall DA. Whole scalp resting state EEG of oscillatory brain activity shows no parametric relationship with psychoacoustic and psychosocial assessment of tinnitus: A repeated measures study. Hear Res. 2016 Jan;331:101-8. doi: 10.1016/j.heares.2015.11.003. Epub 2015 Nov 14. PMID 26584760
- [Background] Fackrell K, Hall DA, Barry JG, Hoare DJ. Response to Letter: Psychometric properties of the Tinnitus Functional Index (TFI): Assessment in a UK research volunteer population. Hear Res. 2016 May;335:237-238. doi: 10.1016/j.heares.2016.03.014. Epub 2016 Mar 30. No abstract available. PMID 27039256
- [Derived] Hall DA, Pierzycki RH, Thomas H, Greenberg D, Sereda M, Hoare DJ. Systematic Evaluation of the T30 Neurostimulator Treatment for Tinnitus: A Double-Blind Randomised Placebo-Controlled Trial with Open-Label Extension. Brain Sci. 2022 Feb 26;12(3):317. doi: 10.3390/brainsci12030317. PMID 35326273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient first visit, 28 May 2012
  Last patient last visit, 26 February 2014
Pre-assignment Details: 217 screen fails: Ménière(6), neuroma(2), TMJ(3), hearing loss(2), new hearing-aid user(11), recent hearing-aid adjustments(2), severe anxiety(4), severe depression(5), pulsatile TI(7), somatic TI(17), intermittent TI(7), slight TI(35), catastrophic TI(6), pitch match not possible(7), pitch out of fitting range(56), prescription tones inaudible(47)
Groups:
- CR Neuromodulation: Acoustic Co-ordinated Reset (CR) Neuromodulation includes an ear level device which delivers patterned sound stimulation. Participants were asked to wear the device for 4-6 hours per day (0-12 weeks) and for at least 4 hours daily (12-36 weeks)
  The experimental arm received the intervention in a double-blind RCT (0-12 weeks), with the device fitted according to audiologist training given by the manufacturer/funder. An individually specified sound stimulation algorithm is hypothesised to interrupt tinnitus generating activity in the brain.
  After the first 12 weeks, the participants entered into the open-label extension (unblinded, 12-36 weeks) in which they continued with the same experimental intervention.
- Tinnitus Masking: The active control group had the same ear level device which delivers patterned sound stimulation. Participants were asked to wear the device for 4-6 hours per day (0-36 weeks).
  The active comparator group received the intervention in a double-blind RCT (0-12 weeks). They received the same device as the treatment group but the sound stimulation was determined according to an algorithm predicted not to break up tinnitus generating activity in the brain. The device may have a tinnitus masking effect in the active comparator group.
  After the first 12 weeks, the participants entered into the open-label extension (unblinded, 12-36 weeks) in which they received the verum experimental intervention.
Period: Double-blind (0-12 Weeks)
Arm/Group | CR Neuromodulation | Tinnitus Masking
Started | 50 | 50
Completed | 44 | 48
Not Completed | 6 | 2
Not completed — Dominant pitch match not possible | 0 | 1
Not completed — Pitch shifted out of fitting range | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 2 | 0
Period: Open Label Extension (12-36 Weeks)
Arm/Group | CR Neuromodulation | Tinnitus Masking
Started | 44 | 48
Completed | 33 | 35
Not Completed | 11 | 13
Not completed — Pitch shifted out of fitting range | 1 | 1
Not completed — Prescription adjusted: tones inaudible | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 6 | 8
Not completed — Adverse Event | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- CR Neuromodulation; Tinnitus Masking: see Protocol section for details
- Total: Total of all reporting groups
Arm/Group | CR Neuromodulation | Tinnitus Masking | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (11.3) | 51.8 (12.2) | 50.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 37 | 54
  Male | 33 | 13 | 46
Hearing level (better ear) [Mean (Standard Deviation); unit: decibel hearing level (dB HL)] — Hearing level is measured by the pure tone audiometric threshold measures, averaged across four frequencies (0.5,1,2,and 4 kHz). Higher number equates to higher hearing thresholds (hearing worse).
  decibel hearing level (dB HL) | 13.1 (10.2) | 14.3 (12.0) | 13.7 (11.2)
Hearing level (worse ear) [Mean (Standard Deviation); unit: decibel hearing level (dB HL)] — Hearing level is measured by the pure tone audiometric threshold measures, averaged across four frequencies (0.5,1,2,and 4 kHz). Higher number equates to higher hearing thresholds (hearing worse).
  decibel hearing level (dB HL) | 18.5 (12.4) | 18.7 (12.4) | 18.6 (12.3)
Tinnitus Handicap Inventory [Mean (Standard Deviation); unit: units on a scale] — Multi-item questionnaire measure of tinnitus severity. Global score (0-100 scale). Higher score indicates greater tinnitus handicap.
  units on a scale | 40.0 (17.4) | 40.9 (15.8) | 40.2 (16.4)
Beck Anxiety Inventory [Mean (Standard Deviation); unit: units on a scale] — Global score (0-63 scale). Higher score indicates more anxiety.
  units on a scale | 4.7 (4.7) | 5.4 (6.6) | 5.1 (5.7)
Beck Depression Inventory [Mean (Standard Deviation); unit: units on a scale] — Multi-item questionnaire measure of depression symptomatology. Global score (0-63 scale). Higher score indicates greater severity of depression.
  units on a scale | 8.7 (6.4) | 9.0 (7.3) | 8.7 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Tinnitus Handicap Questionnaire (THQ)
Description: Change in the global score on a 27 item, multi-attribute questionnaire measure of the functional impact of tinnitus (0-100 scale). Change was computed as 'visit 2' - 'visit 6' and so a positive change score indicates a reduction of tinnitus symptoms.
Time Frame: Baseline (visit 2) and 12 weeks (visit 6)
Population: We have analyzed both complete case and multiple imputed data for the mean change in global THQ score from baseline (visit 2) to 12 weeks (visit 6). Here we report complete case data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR Neuromodulation | Tinnitus Masking
Number analyzed (Participants) | 42 | 44
units on a scale | 3.75 (13.29) | 4.02 (9.56)

2. Secondary Outcome: Tinnitus Handicap Inventory (THI)
Description: Change in the global score on a 25 item, multi-attribute questionnaire measure of the functional impact of tinnitus (0-100 scale). Change was computed as 'visit 2' - 'visit 6' and so a positive change score indicates a reduction of tinnitus symptoms.
Time Frame: Baseline (visit 2) and 12 weeks (visit 6)
Population: We have analyzed both complete case and multiple imputed data for the mean change in global THI score from baseline (visit 2) to 12 weeks (visit 6). Here we report complete case data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR Neuromodulation | Tinnitus Masking
Number analyzed (Participants) | 43 | 45
units on a scale | 2.84 (14.89) | 1.64 (10.81)

3. Secondary Outcome: Tinnitus Functional Index (TFI)
Description: as for outcome 2
Time Frame: Baseline (visit 2) and 12 weeks (visit 6)
Population: We have analyzed both complete case and multiple imputed data for the mean change in global TFI score from baseline (visit 2) to 12 weeks (visit 6). Here we report complete case data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR Neuromodulation | Tinnitus Masking
Number analyzed (Participants) | 43 | 45
units on a scale | 2.38 (19.70) | 4.45 (14.85)

4. Secondary Outcome: World Health Organization Quality of Life Questionnaire (WHOQOL-BREF)
Description: The WHOQOL-BREF is a 26-item, multi-attribute questionnaire measure of health related quality of life. Outcome was measured as a change on Question 1: 'How would you rate your quality of life (over the past 4 weeks)?' There are 5 response options (Very poor=1; Poor=2; Neither poor nor good=3; Good=4; Very good=5). Change was computed as 'visit 2' - 'visit 6' and so a positive change score indicates a reduction in self-perceived quality of life.
Time Frame: Baseline (visit 2) and 12 weeks (visit 6)
Population: We have analyzed both complete case and multiple imputed data for the mean change in Q1 score from baseline (visit 2) to 12 weeks (visit 6). Here we report complete case data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR Neuromodulation | Tinnitus Masking
Number analyzed (Participants) | 43 | 45
units on a scale | -0.21 (0.64) | -0.11 (0.61)

5. Secondary Outcome: Percent Change From Baseline in Normalized Oscillatory Power in the Delta Brainwave Pattern as Measured by Electroencephalography (EEG)
Description: Non-invasive recording to measure rhythmic patterns of spontaneous brain activity at rest. An a priori hypothesis targeted normalized delta rhythm. Band powers were calculated as percent change in delta brainwave pattern relative to change in total (1-90 Hz) EEG band. Comparison made between 'visit 2' and 'visit 6'.
  We used a Neuroscan system (SynAmps2 model 8050, Compumedics Neuroscan, Charlotte, NC, USA) and custom cap with 66 equidistant scalp electrodes (Easycap, GmbH, Germany). A central frontal electrode was used as ground and a nose-tip electrode as reference. Electrode impedances were maintained at 5 kΩ prior to recordings. Recording was done with an offline filter of 0.5 to 200 Hz pass-band and 1 kHz sampling rate. Recording was over a continuous 10-minute period. Participants were seated in a quiet, darkened soundproof booth and were instructed to relax, keep eyes open and fix gaze on a marker point.
Time Frame: Baseline (visit 2) and 12 weeks (visit 6)
Population: The EEG assessment was offered only to the first 50 participants enrolled at the Nottingham site. We have analyzed only complete case data for the mean change in delta band power from baseline (visit 2) to 12 weeks (visit 6).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | CR Neuromodulation | Tinnitus Masking
Number analyzed (Participants) | 20 | 22
Percent change | 0.001 (0.01) | 0.004 (0.013)

6. Secondary Outcome: Tinnitus Handicap Questionnaire (THQ)
Description: Change in the global score on a 27 item, multi-attribute questionnaire measure of the functional impact of tinnitus (0-100 scale). Change was computed as 'visit 2' - 'visit 10' and so a positive change score indicates a reduction of tinnitus symptoms.
Time Frame: Baseline (visit 2) and 36 weeks (visit 10)
Population: We have analyzed both complete case and multiple imputed data for the mean change in global THQ score from baseline (visit 2) to 36 weeks (visit 10). Here we report complete case data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CR Neuromodulation: The treatment group were unblinded at 12 weeks and then continued to receive the same experimental intervention. At 36 weeks, this group had therefore received active treatment (0-36 weeks).
- Tinnitus Masking: The active comparator group were unblinded at 12 weeks and the device algorithm was reprogrammed in the same way as the experimental intervention. At 36 weeks, this group had therefore received a mixture of placebo (0-12 weeks) and active treatment (12-36 weeks).
Arm/Group | CR Neuromodulation | Tinnitus Masking
Number analyzed (Participants) | 30 | 33
units on a scale | 5.41 (15.64) | 6.01 (10.52)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected across the 36 weeks.
Description: The definition of an adverse event in the context of this study is: (1) since wearing the ear-level device tinnitus intrusiveness increased and made the condition unbearable, (2) a disease or symptoms (unrelated to tinnitus) that was present at baseline and wosened following the start of the study.
Groups:
- Acoustic CR Neuromodulation; Tinnitus Masking: see Protocol section for details
Arm/Group | Acoustic CR Neuromodulation | Tinnitus Masking
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 4/50 | 3/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acoustic CR Neuromodulation (N=50) | Tinnitus Masking (N=50)
Tinnitus worsened (Ear and labyrinth disorders) | 4 (4) | 3 (3) — In Acoustic CR Neuromodulation group AE reported by 2 participants during 12 week RCT phase, and 2 participants in the LTE phase (weeks 13 to 36). In the Tinnitus Masking group AE reported by 3 participants in the LTE phase (after crossover).

LIMITATIONS AND CAVEATS:
Clinical Trial Protocol inadequately specified, particularly (i) device fitting, (ii) tolerance for pitch matching shifts and (iii) monitoring research audiologists after training. Specification of placebo algorithm is not evidenced by published data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The manufacturer acknowledges and accepts the right of the investigator to publish the results of the research, however, the Investigator shall send a draft manuscript of the publication or abstract of the study findings to the manufacturer 30 days in advance of submission to a scientific journal for approval. Adaptive Neuromodulation GmbH was the manufacturer at the start of the trial, subsequently passing to NeuroTherapies Reset (Brook Henderson Group) during open-label extension.